CLINICAL TRIAL: NCT04168775
Title: A Single Center, Open Label, Prospective Study Measuring Proportion of Patients With Suboptimal Peak Inspiratory Flow Rate (sPIFR) Over 24 Weeks in an Ambulatory Setting Among Moderate to Very Severe COPD Patients
Brief Title: Peak Inspiratory Flow Rates in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-0450
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: COPD
Keywords: peak inspiratory flow rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Home PIFR monitoring (Other): Measurement of PIFR using the InCheck Dial® device and quantification of respiratory symptoms and COPD exacerbations using standardized questionnaires in the patient's home setting and during research visits in the clinic setting
  Interventions: Device: Home PIFR monitoring with InCheck Dial

INTERVENTIONS:
Device: Home PIFR monitoring with InCheck Dial — The In-Check G16 DIAL® (Alliance Tech Medical, Granbury TX) is a simple hand-held device that measures PIFR via a brief inspiratory maneuver.

SUMMARY:
Recent studies have reported that some Chronic Obstructive Pulmonary Disease (COPD) patients may have a suboptimal ability to generate a sufficient inspiratory effort to achieve adequate lung delivery of inhaled medications through dry powder inhalers. Sparse data is available about the inspiratory capacity of these patients in the home setting, whether clinically stable or when experiencing worsened respiratory symptoms outside the acute care setting. This study is undertaken to better understand the proportion of patients with suboptimal peak inspiratory flow rate (sPIFR) measurements amongst COPD patients receiving dry powder inhaler(s) (DPI) in the ambulatory setting. Further, the study will characterize PIFR over time, the variability of PIFR measurements, and the associations with potential predictors (demographics, clinical, Patient-Reported Outcomes (PRO), body position, and device) as well as exacerbations frequency and change in PIFR around period of exacerbation.

DETAILED DESCRIPTION:
Recent studies have reported that some COPD patients may have a suboptimal ability to generate a sufficient inspiratory effort to achieve adequate lung delivery of inhaled medications through dry powder inhalers. Sparse data is available about the inspiratory capacity of these patients in the home setting, whether clinically stable or when experiencing worsened respiratory symptoms outside the acute care setting. This study is undertaking this study to better understand the proportion of patients with suboptimal peak inspiratory flow rate (sPIFR) measurements amongst COPD patients receiving dry powder inhaler(s) (DPI) in the ambulatory setting. Further, the study will characterize PIFR over time, the variability of PIFR measurements, and the associations with potential predictors (demographics, clinical, PRO, body position, and device) as well as exacerbations frequency and change in PIFR around period of exacerbation. To complete these aims, 120 participants will be enrolled in a 6 month study to perform PIFR measurements and respiratory questionnaires at home.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years-old
* Spirometry-confirmed diagnosis of COPD (FEV1/FVC <0.70)
* Global initiative for Chronic Obstructive Lung Disease (GOLD) II-IV based on spirometry results
* COPD Assessment Test (CAT) score > 10
* For high resistance DPI, baseline PIFR < 90 L/min (InCheck DIAL®) and >=30 L/min; for medium resistance DPI, PIFR ≤ 90 L/min (InCheck DIAL®) and >=60 L/min. Handihaler is a high resistance DPI. Examples of medium resistance DPI: Anoro, Incruse, Breo Ellipta®, Advair® Diskus® DP or Wixela® Inhub®
* History of smoking tobacco products > 10 pack years
* Prescribed at least one daily maintenance DPI with no change in prescription within the four weeks prior to the Enrollment Visit
* One or more exacerbations of COPD requiring systemic corticosteroids within last 2 years

Exclusion Criteria:

* Inability to demonstrate proper technique for the InCheck DIAL® device
* Inability to achieve minimum PIFR for prescribed DPI(s) at screening/enrollment visit (< 30 L/min for e.g., Handihaler® (High resistance DPI), < 60 L/min for Ellipta® (Medium resistance DPI))
* Inability to perform spirometry to meet American Thoracic Society standards
* Neuromuscular disease associated with weakness
* Any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study.
* Pneumothorax within the past 4 weeks
* For those participants who will require spirometry (i.e., if they have not had it within the past 3 months): Participants who present with a myocardial infarction or eye, chest or abdominal surgery within six weeks of baseline can be rescreened after the six week window has passed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Drummond, MD, Principal Investigator — University of North Carolina, Chapel Hill; Ashley Henderson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pleasants RA, Shaikh A, Henderson AG, Bayer V, Drummond MB. Changes in Peak Inspiratory Flow After Acute Bronchodilation: An Observational Study of Patients with Stable Chronic Obstructive Pulmonary Disease. J Aerosol Med Pulm Drug Deliv. 2024 Aug;37(4):171-179. doi: 10.1089/jamp.2023.0045. Epub 2024 May 29. PMID 38814000
- [Derived] Pleasants RA, Henderson AG, Bayer V, Shaikh A, Drummond MB. Effect on Physical Position of Peak Inspiratory Flow in Stable COPD: An Observational Study. Chronic Obstr Pulm Dis. 2024 Mar 26;11(2):174-186. doi: 10.15326/jcopdf.2023.0460. PMID 38236166

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home PIFR Monitoring
Started | 80
Completed | 75
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Home PIFR Monitoring
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Suboptimal PIFR
Description: The occurrence of suboptimal Peak Inspiratory Flow Rate (sPIFR) over 24 weeks. sPIFR will be defined as any two consecutive measurements on different days below the optimal threshold for any prescribed DPI (e.g.,<30 L/min for Handihaler® (High resistance DPI), <60 L/min for Ellipta® (Medium resistance DPI))
Time Frame: 24 weeks
Population: Data are reported for all participants who contributed at least 2 consecutive PIFR measurements on different days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Home PIFR Monitoring
Number analyzed (Participants) | 75
percentage of participants | 22.7 [13.8 to 33.8]

ADVERSE EVENTS:
Time Frame: From Screening when participants signed Informed Consent through last completed study visit, a total of up to approximately 6 months.
Arm/Group | Home PIFR Monitoring
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 22/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home PIFR Monitoring (N=80)
COPD Exacerbation leading to Hospitalization (Respiratory, thoracic and mediastinal disorders) | 22 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04168775/Prot_SAP_000.pdf